CLINICAL TRIAL: NCT01483677
Title: Is Nintendo Wii a More Suitable Video Game Platform Than Playstation 2 for Enhancing Laparoscopic Skills?
Brief Title: Comparison Study of the Nintendo Wii Versus Playstation2 in Enhancing Laparoscopic Skills
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 023-10
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Laparoscopy Skills
Keywords: Laparoscopy; video games; Nintendo Wii; Playstation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nintendo Wii (Experimental): Subjects in this arm of the study play a game (Boomblox) on the Nintendo Wii for 30 minutes.
  Interventions: Other: Nintendo Wii
- Playstation2 (Active Comparator): Subjects in this arm of the study play a game (Time Crisis 2) on the Playstation 2 for 30 minutes.
  Interventions: Other: Playstation 2

INTERVENTIONS:
Other: Nintendo Wii — Subjects played the game Boomblox for 30 continuous minutes on the Nintendo Wii.
  Other Names: Boomblox
  Arms: Nintendo Wii
Other: Playstation 2 — Subjects played the game Time Crisis2 on the Playstation2 for 30 continuous minutes.
  Other Names: Time Crisis
  Arms: Playstation2

SUMMARY:
The investigators believe that subjects who practice on the Nintendo Wii will improve their laparoscopic skills more than those who practice on the Playstation2.

DETAILED DESCRIPTION:
Video game experience, whether past or current, have correlated with better laparoscopy skills. Those studies were conducted using traditional game controllers. The relatively new Nintendo Wii uses a novel set of mechanics which allows for more realistic representation of player generated movements. We aim to study if the unique mechanics of the Wii can improve laparoscopy skills better than a traditional video game (Playstation 2).

ELIGIBILITY:
Inclusion Criteria:

* Medical Student, Resident or Attending physician at the Beth Israel Medical center.

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Difference in the change in box trainer scores between the Wii and Playstation2 groups. | 60 minutes
  After completion of the pretest, subjects are given a 10 minute break, 30 minutes of video game play, a 10 minute break, and 10 minutes to complete the post test.

SECONDARY OUTCOMES:
Change between pretest and post test scores in the Wii group. | 60 minutes.
  After completion of the pretest, subjects are given a 10 minute break, 30 minutes of video game play, a 10 minute break, and 10 minutes to complete the post test.
Change between pretest and posttest scores for the Playstation2 group | 60 minutes
  After completion of the pretest, subjects are given a 10 minute break, 30 minutes of video game play, a 10 minute break, and 10 minutes to complete the post test.

CONTACTS AND LOCATIONS:
Overall Officials: Rujin Ju, M.D., Principal Investigator — Beth Israel Medical Center; Karen C Wang, M.D., Study Chair — Brigham and Women's Hospital
Locations (1):
- Beth Israel Medical Center of The Albert Einstein College of Medicine, New York, New York, United States

REFERENCES:
- [Background] Derossis AM, Bothwell J, Sigman HH, Fried GM. The effect of practice on performance in a laparoscopic simulator. Surg Endosc. 1998 Sep;12(9):1117-20. doi: 10.1007/s004649900796. PMID 9716763
- [Background] Rosser JC Jr, Lynch PJ, Cuddihy L, Gentile DA, Klonsky J, Merrell R. The impact of video games on training surgeons in the 21st century. Arch Surg. 2007 Feb;142(2):181-6; discusssion 186. doi: 10.1001/archsurg.142.2.181. PMID 17309970
- [Background] Smith CD, Farrell TM, McNatt SS, Metreveli RE. Assessing laparoscopic manipulative skills. Am J Surg. 2001 Jun;181(6):547-50. doi: 10.1016/s0002-9610(01)00639-0. PMID 11513783
- [Background] Lewis TM, Aggarwal R, Rajaretnam N, Grantcharov TP, Darzi A. Training in surgical oncology - the role of VR simulation. Surg Oncol. 2011 Sep;20(3):134-9. doi: 10.1016/j.suronc.2011.04.005. Epub 2011 May 24. PMID 21605972
- [Background] Munz Y, Kumar BD, Moorthy K, Bann S, Darzi A. Laparoscopic virtual reality and box trainers: is one superior to the other? Surg Endosc. 2004 Mar;18(3):485-94. doi: 10.1007/s00464-003-9043-7. Epub 2004 Feb 2. PMID 14752633
- See also: Mechanical engineering aspect of Wii — http://www.engeneration.imeche.org/